CLINICAL TRIAL: NCT03090009
Title: The Use of Non-Steroidal Anti-Inflammatory Drugs as a Tool of Positive Change in Peri-Implants Mucositis Microbiome
Brief Title: Microbiome Shift in Peri-mucositis by Anti-inflammatory Drugs
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Polak David (Other)
Responsible Party: Sponsor-Investigator, Polak David, Principal Investigator, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0674-16-HMO
Record Dates: First submitted 2017-03-02; First posted 2017-03-24 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Peri-implant Mucositis
Keywords: Peri-implant Mucositis; NSAID; Microbiome; 16s Ribosomal Pyro-sequencing
MeSH Terms: interventions — Flurbiprofen; strepfen

STUDY DESIGN:
Intervention Model Description: The study design is random controlled double blind clinical trial
Who Masked: Participant, Investigator
Masking Description: Both patient and investigator will blinded to the identity of the medication given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flurbiprofen (Active Comparator): Flurbiprofen 100 mg bid.
  Interventions: Drug: Flurbiprofen
- Placebo (Placebo Comparator): Placebo taken bid
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Flurbiprofen — 100 mg twice a day for 14 days
  Other Names: Ansaid; Strepfen; Ocufen
  Arms: Flurbiprofen
Drug: Placebo Oral Tablet — placebo group
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Dental implants are often used to replace missing teeth. In fact, in the US over 700,000 implants are places every year and over 2 million implants are places world wide. Peri-implant mucositis in an inflammatory condition affecting dental implants and is recognized as a risk factor for peri-implantitis (a condition affecting the bone around implants and eventually leading to implant loss). The prevalence of Peri-implant Mucositis has been reported in the literature to range from 50-90% whereas the prevalence of Peri-implantitis has been reported as high as 20%. it is commonly believed that a dysbiotic microbiome is the primary cause for these conditions.

The inflammatory burden around diseased implants creates a high-protein environment which is necessary for the survival of pathogenic bacteria. It is logical, therefore, that reducing inflammation by Non Steroidal Anti-Inflammatory Drugs (NSAIDs) may create a shift in the dysbiotic microbiome to a symbiotic microbiome. The aim of the current study is to test the effects of oral NSAIDs on the peri-implant microbiome.

DETAILED DESCRIPTION:
Inflammation around dental implants has been defined as Peri-implant mucositis and Peri-implantitis . Peri-implant mucositis is a localized inflammation limited to the mucosal tissue surrounding the implant whereas peri-implantitis has advanced to the bone surrounding the implant as well. The prevalence of Peri-implant Mucositis has been reported in the literature to range from 50-90% whereas the prevalence of Peri-implantitis has been reported as high as 20%. Due to the fact that there are many similarities in the clinical manifestations of infection in the gingiva and peri-implant mucosal tissue, studies attempted to compare the microbial characteristics around teeth to that found around implants. Emerging data suggests that the microbiome around infected teeth has some similarities and dissimilarities to peri-implant infection. Such differences may stem from different inflammatory characteristics as well as the presence of a non-vital foreign material (the dental implant) in the area. Some of the known pathogenic strains identified in the peri-implant sulcus are anaerobic a-saccharolytic bacteria, which feed off the adjacent tissue inflammatory exudate. Logically, attenuation of the inflammation would deprive the nearby bacteria of nourishment needed to sustain their growth.

The use of non-steroidal anti-inflammatory drugs (NSAID) to control chronic inflammatory disease has been used extensively in medicine. Its action of blocking cyclooxygenase inflammatory pathway and in-effect blocking the production of Prostaglandin-E2 (PGE2) has led to its use with general pain control as well as its long term use in the treatment of tissue inflammation and pain caused by rheumatoid arthritis or osteoarthritis, tendinitis and bursitis.

Offenbacher et al. as early as in 1981 discovered that patients with periodontitis had significantly higher levels of PGE2 in the sulcular fluid between gingiva and the tooth (GCF) . In a follow up study over a period of 18-36 months, Offenbacher observed that patients who had exhibited periodontal attachment loss had significantly higher levels of PGE2. This led Williams et al. to study the effects of Flurbiprofen, a phenylalkanoic derivative family of of non-steroidal anti-inflammatory drugs, on naturally occurring periodontal disease in an animal model over a period of 12 months. The study demonstrated decreases in alveolar bone loss in flurprofen treated animals at 3, 6 , 9 and 12 months. William et al then followed with a clinical trial where 44 patients who self administered peroral flurbiprofen twice daily for a period of 24 months. The study reported severely depressed bone loss rates over the period of the trial and as early as 6 months after administration of flurbiprofen that continued over the length of the trial. Other studied the drugs effect on other more aggressive forms of the disease with similar results . These results have been duplicated around implants as well. Jeffcoat et al demonstrated that oral intake flurbiprofen helped reduce bone loss around implants in the first year of service. Reddy similarly demonstrated with use of digital subtraction radiography, flurbiprofen taken orally was able to help increase bone density and apposition around implants after just 4 months.

The positive effect of systemic antibiotics and as well topical anti microbials on the pathogenic bacteria in the gingiva sulcus and peri-implant crevice has been well documented and is indisputable. The removal of these bacteria has helped promote tissue health. Similar results have been documented around implants as well. However more recently the reverse approach to disease control has gained popularity. Instead of trying just to reduce the bacterial challenge through antimicrobial/antibiotic therapy, modulating the host response to decrease the inflammatory destruction of the tissue, could be a more efficient and effective way of controlling the disease In decreasing the inflammatory environment, the pathogenic bacteria feeding off the inflammatory exudate would be greatly decreased, effecting a major change in the microbiome. To date nobody has characterized this change.

The purpose of the study is to test the effects of oral NSAIDS on the peri-implant microbiome. Also, clinical parameters will be tested for correlation with the microbial findings.

Methods:

The study design is random controlled double blind clinical trial. Patients visiting the graduate periodontal clinic at the Hadassah Medical Center will be examined for eligibility for the study. Implants with peri-implant mucositis (clinical signs of inflammation without radiographically bone loss) will be included. Patients (n=50) will undergo clinical examination (which will include probing depths, presence or absence of suppuration and bleeding on probing) and sampling of the subgingival bacterial deposits using a perio-strip. Patients will be randomly assigned to the experimental flurbiprofen group (100 mg bid) or placebo group (n=25 for each group). Drug consumption will be set for the duration of 2 weeks. At the end of drug intake period (day 14) and two weeks afterwards (day 28) all subjects will be re-examined, which will include a new clinical exam and sampling of the subgingival bacterial deposits. The microbiological samples will be analyzed using 16s Ribosomal Pyro-sequencing. The microbiome profile of the Flurbiprofen group before and after treatment and two weeks post-treatment will be compared. as well as the microbiome from the placebo group compared with the Flurbiprofen group. Statistical differences will be evaluated using ANOVA with Bonferroni correction. Correlation between the clinical parameters and microbiological parameters will be tested using Pearson correlation.

Significance:

The study asks the question whether the use of a well-known NSAID that had proven beneficial effects in maintaining the mucosal tissue integrity around implants and help control and prevent peri-implant inflammation. Studies have shown that implants placed 5 years previously will most likely have some form of peri-implant mucositis . Just as gingivitis can lead to periodontal disease, Peri-implant mucositis can lead to peri-implantitis a more destructive inflammatory disease that puts implant survival in jeopardy. Therefore, a drug that can limit the amount of destructive bacteria around the implant can be a very effective non-invasive method of treatment. Additionally with the use of a more comprehensive taxonomical identification of the peri-implant micro-genome, there will be a better understanding of the bacterial role in the destructive process associated with peri-implant inflammation

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Peri-implant Mucositis

Exclusion Criteria:

* hypersensitivity to or intolerance of Flurbiprofen or NSAIDs
* peptic ulcer
* pregnancy
* smoking
* diabetes mellitus
* having taken any antibiotic drug within the previous 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in the Microbiome | 28 days
  The microbiome profile of the Flurbiprofen group before treatment (base line) and after treatment (day 14) and two weeks post-treatment (day 28) will be compared, as well as the microbiome of the placebo group. data will be pooled and analysed as absolute number of any microbe within the tested biofilms. Measures of change will be set as 14d vs. baseline and 28 day vs. baseline.

SECONDARY OUTCOMES:
change in periodontal probing depth | 28 days
  change in probing sulcular depth around implants
change in bleeding on probing | 28 days
  change in bleeding on probing in the peri-implant sulcus
change in Suppuration | 28 days
  change in presence or absence in the peri-implant sulcus

CONTACTS AND LOCATIONS:
Overall Officials: David Polak, DMD PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paquette DW, Williams RC. Modulation of host inflammatory mediators as a treatment strategy for periodontal diseases. Periodontol 2000. 2000 Oct;24:239-52. doi: 10.1034/j.1600-0757.2000.2240112.x. PMID 11276870
- [Background] Jeffcoat MK, Reddy MS, Wang IC, Meuninghoff LA, Farmer JB, Koth DL. The effect of systemic flurbiprofen on bone supporting dental implants. J Am Dent Assoc. 1995 Mar;126(3):305-11; quiz 346-7. doi: 10.14219/jada.archive.1995.0173. PMID 7646652